CLINICAL TRIAL: NCT06755970
Title: The Effect of the ICOUGH Bundle Applied Under Nurse Leadership on Pain and Nausea After Laparoscopic Cholecystectomy: a Randomized Controlled Study
Brief Title: ICOUGH Bundle and Postoperative Pain and Nausea After Laparoscopic Cholecystectomy
Acronym: ICOUGHBundle
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, MERVE KAYA, pricipal investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AtaturkUnıversty
Record Dates: First submitted 2024-12-18; First posted 2025-01-01 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-12

CONDITIONS: Laparoscopic Cholecystectomy; Pain; ICOUGH; NAUSEA
Keywords: Pain; Laparoscopic cholecystectomy; Nausea
MeSH Terms: conditions — Pain; Nausea

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Grup 1 (Experimental): The ICOUGH care bundle will be applied to this group.
  Interventions: Procedure: ICOUGH
- Control grup: Grup 2 (No Intervention): The ICOUGH care bundle will not be applied to this group.

INTERVENTIONS:
Procedure: ICOUGH — After the patient has recovered from postoperative anesthesia and their hemodynamic values have stabilized, the ICOUGH bundle applications mentioned above will be carried out. The patient's pain and nausea levels will be recorded for a period of 48 hours.
  Postoperative pain and nausea will be assessed with the help of data collectors, using a numerical rating scale at 2, 4, 8, 12, 24, and 48 hours after surgery.
  Considering that postoperative respiratory complications are relatively common and costly, various studies have been conducted to explore ways to reduce the risk of their occurrence. One of these protocols is the ICOUGH bundle, which stands for Incentive Spirometry, Coughing and Deep Breathing, Oral Care, Patient Understanding of the Interventions, Getting Out of Bed, and Head of Bed Elevation.
  Arms: Experimental: Grup 1

SUMMARY:
This study will use a randomized controlled experimental research design. The population of the study will consist of all adult patients who undergo laparoscopic cholecystectomy at the General Surgery Clinic of Atatürk University Research Hospital between December 2024 and September 2025. The data will be collected using a Descriptive Information Form and the Visual Analogue Scale. The research has received institutional approval and ethics committee approval. The study will be conducted with collaboration from healthcare professionals in the clinic after they have been informed. Patients who meet the inclusion criteria will be invited to participate in the study after being approached one day before surgery. Oral and written consent will be obtained from those who volunteer and agree to participate. The data will be analyzed using SPSS for Windows 22 software.

DETAILED DESCRIPTION:
Post-laparoscopic cholecystectomy, patients may experience pain at the incision site, internal organ pain, and shoulder pain. Shoulder pain occurs due to the irritation of the diaphragm peritoneum by dissolved CO2 gas, causing the diaphragm to stretch, which stimulates the phrenic nerve and results in shoulder pain in these patients. This shoulder pain is typically felt up to 72 hours or three days after surgery.

Shoulder pain in these patients is typically felt for up to 72 hours or three days after surgery. Pneumoperitoneum during laparoscopy can also produce vagal stimulation, which can lead to nausea and vomiting. In this context, the removal of CO2 is essential for managing post-laparoscopic cholecystectomy CO2-related pain.

Given the relatively common and costly occurrence of postoperative respiratory complications, various protocols have been used to reduce the risk of these complications. One such protocol is the ICOUGH (Incentive spirometry, Coughing and deep breathing, Oral care, Patient understanding of the interventions, Getting out of bed and Head of bed elevation) bundle, developed by the Boston University School of Medicine in 2012 to reduce postoperative respiratory complications. This respiratory care bundle improves oxygenation and CO2 elimination, thus increasing the patient's recovery rate, reducing the amount of analgesics used, and shortening the time to return to daily activities.

The ICOUGH bundle, which is among the important independent responsibilities of perioperative nurses, helps reduce shoulder pain and accelerate postoperative recovery by increasing CO2 elimination and oxygenation. The use of non-pharmacological methods for pain relief in the postoperative period strengthens the nurse's role in pain management. The aim of this study is to determine the effects of the ICOUGH bundle on shoulder pain, abdominal pain, and nausea after laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Those who agree to participate in the study and volunteer
* Aged 18 and above
* Undergoing laparoscopic cholecystectomy surgery under general anesthesia
* Those without physical or mental disabilities, limitations, or conditions that would prevent them from performing respiratory exercises (such as the use of medications affecting respiration, conditions requiring oxygen therapy, etc.)
* Those whose cognitive level is suitable for the application of scales
* Patients without communication problems will be included in the study

Exclusion Criteria:

* Those whose hemodynamic values are not stable after the surgical intervention
* Those who develop any complications such as severe bleeding, nausea, vomiting, etc., after surgery
* Patients with acute or chronic lung diseases
* Patients who voluntarily wish to withdraw from the study will not be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 2nd hour after surgery
  Patients are asked to rate their pain level on a horizontal line between 0 and 10. 0 represents no pain, and 10 represents unbearable pain. Due to its simplicity, validity, and reliability, it is used as the most suitable tool to assess pain intensity. It can be used to evaluate both pain and nausea.
Visual Analog Scale (VAS) | 4nd hour after surgery
  Patients are asked to rate their pain level on a horizontal line between 0 and 10. 0 represents no pain, and 10 represents unbearable pain. Due to its simplicity, validity, and reliability, it is used as the most suitable tool to assess pain intensity. It can be used to evaluate both pain and nausea.
Visual Analog Scale (VAS) | 8nd hour after surgery
  Patients are asked to rate their pain level on a horizontal line between 0 and 10. 0 represents no pain, and 10 represents unbearable pain. Due to its simplicity, validity, and reliability, it is used as the most suitable tool to assess pain intensity. It can be used to evaluate both pain and nausea.
Visual Analog Scale (VAS) | 12nd hour after surgery
  Patients are asked to rate their pain level on a horizontal line between 0 and 10. 0 represents no pain, and 10 represents unbearable pain. Due to its simplicity, validity, and reliability, it is used as the most suitable tool to assess pain intensity. It can be used to evaluate both pain and nausea.
Visual Analog Scale (VAS) | 24nd hour after surgery
  Patients are asked to rate their pain level on a horizontal line between 0 and 10. 0 represents no pain, and 10 represents unbearable pain. Due to its simplicity, validity, and reliability, it is used as the most suitable tool to assess pain intensity. It can be used to evaluate both pain and nausea.

IPD SHARING:
Plan to Share IPD: No